CLINICAL TRIAL: NCT05148611
Title: Application Registration Study of ILE in Patients With Acute Poisoning
Acronym: ILE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); People's Hospital of Deyang City (Unknown); Binzhou Medical University (Other); People's Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-3185D
Record Dates: First submitted 2021-11-01; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-09

CONDITIONS: Acute Poisoning
Keywords: Acute poisoning; intravenous lipid emulsion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Take the patient's blood for general laboratory tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators aimed to study the effect of ILE in the treatment of acute fat-soluble substance poisoning,to further clarify the relevant mechanism of ILE in the treatment of fat-soluble drug poisoning,to standardize the relevant procedures of ILE detoxification treatment and further explore the adverse reactions and coping strategies of ILE treatment.

DETAILED DESCRIPTION:
Fat-soluble drugs refer to drugs that are insoluble in water but soluble in fats and organic solvents such as carbon tetrachloride, glycerol, oils and other organic solvents. They can fuse with the phospholipid bilayer of cell membranes, are easily absorbed, and are easier to pass compared to water-soluble drugs. It is metabolized by the liver, and the metabolites are excreted by the kidneys, so it has a high clinical use rate. However, in recent years, due to the improper use of fat-soluble drugs by patients, fat-soluble benzodiazepines sedative and hypnotic drugs, fat-soluble calcium channel blockers and β-blocker drugs, fat-soluble tricyclic drugs have often occurred. Poisoning such as antidepressants poses a serious threat to the lives of patients.In addition, organophosphorus pesticides (fat-soluble) have a high usage rate in China. Severe organophosphorus poisoning can cause multiple organ damages, and delays in treatment can cause disability or even death. Clinical treatment is mainly based on routine gastric lavage and oxygen inhalation. Treatment is the mainstay, combined with medical drugs, hemodialysis, hemoperfusion, etc., and has achieved certain curative effects, but the mortality rate is still high, so it is of great significance to explore safer and more effective treatment methods.Intravenous lipid emulsion (ILE) was originally used to treat overdose of local anesthetics such as bupivacaine, and later also used to treat a variety of other lipophilic drug poisonings. The research on the treatment of ILE is still in the preliminary stage and relatively limited. A systematic review of fat emulsions for the treatment of acute poisoning found that the overall quality of the studies supporting this treatment is low or very low, but the included case reports indicate that fat emulsions are effective against verapamil, beta blockers, and certain Tricyclic antidepressants, bupivacaine, chlorpromazine, and certain antiarrhythmic drugs (eg, flecainide) poisoned patients have certain benefits. ILE may help treat patients who are hemodynamically unstable due to poisoning by these drugs.In view of the fact that the research on the treatment of ILE still needs to be further improved and related adverse reactions need to be further explored related countermeasures, the investigators plan to launch a registration research program related to the application of fat emulsion.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as acute fat-soluble drug and organophosphorus (fat-soluble) pesticide poisoning;
2. Conventional treatment is ineffective, especially for patients with circulatory failure, such as ventricular arrhythmia, shock, cardiac arrest, etc., who need intravenous fat emulsion treatment;
3. Those who are not allergic to fat milk;
4. Sign informed consent.

Exclusion Criteria:

1. Mergers with insufficiency of important organs;
2. Patients with malignant tumors;
3. Severe mental disorder affects the treatment;
4. Those with incomplete clinical data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: According to the indications of ILE in the treatment of poisoning in clinical toxicology, the research objects are divided into the following categories:
  1. Calcium channel blocker poisoning
  2. Beta blocker drug poisoning
  3. Tricyclic antidepressant poisoning
  4. Organophosphorus (fat-soluble) pesticide poisoning, such as: chlorpyrifos, profenofos, diazinon, fenthion, phosphaphos, quinalphos, butylpyrimidin, thiazophos, omethoate, dimethoate Methionine, triazophos, thiomethionine, ethion, sulfoxiphos, imiphos, fosfoxcarb, pyrifoxaphos, hydrocarbophos, phorate, methyl parathion, parasulfur Phosphorus, dichlorvos, pyridoxine, etc.
  5. Local anesthetic poisoning
  6. Poisoning by other fat-soluble substances
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 24 hours
  Patient mortality within 24 hours

SECONDARY OUTCOMES:
Circulatory system | 24 hours
  Circulation stabilization time: including blood pressure stabilization time, disappearance time of malignant arrhythmia, etc.
mortality rate | 1 week and 28 days
  1 week and 28 days patient mortality

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT05148611/Prot_000.pdf
  • Informed Consent Form (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT05148611/ICF_001.pdf